CLINICAL TRIAL: NCT00877344
Title: Better Contraceptive Choices: Immediate vs. Delayed Insertion of Intrauterine Contraception After Second Trimester Abortion
Brief Title: Better Contraceptive Choices: Immediate or Delayed Insertion of IUC After Second Trimester Abortion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Women's Health Research Institute of British Columbia (Other); College of Family Physicians of Canada (Other)
Responsible Party: Principal Investigator, Wendy Norman, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H09-00363
Record Dates: First submitted 2009-04-03; First posted 2009-04-07 (Estimated); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Pregnancy
Keywords: Pregnancy; IUC; abortion; contraception

STUDY DESIGN:
Intervention Model Description: This study uses a drug (levonorgestrel-releasing intrauterine contraception ("Mirena" (R)), but as the study is conducted in Canada the FDA approval is not required. We have approval (a Letter of No Objection) from the Canadian Equivalent Institution: "Health Canada"
Who Masked: Outcomes Assessor
Masking Description: The assessment of outcomes (pregnancy conceived within one year) will be assessed through documentation of pregnancy in health administrative data.
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Immediate insertion of either a LNG-IUC or a Copper T380 IUD after 12-24 week abortion
  Interventions: Procedure: Immediate insertion
- 2 (Experimental): Interval insertion (two to four weeks post abortion) of either a LNG-IUC or a Copper T380 IUD after 12-24 abortion
  Interventions: Procedure: Interval insertion

INTERVENTIONS:
Procedure: Immediate insertion — Immediate timing of insertion for a LNG-IUC OR Copper 380mg T-shaped IUD after an abortion for a gestational age between 12 weeks zero days and 23 weeks 6 days. Immediate insertions occur during the visit for the abortion immediately after the abortion is complete, interval insertions will be scheduled for not earlier than two weeks and not later than four weeks after the abortion.
  Arms: 1
Procedure: Interval insertion — Interval Timing of insertion for a LNG-IUC OR Copper 380mg T-shaped IUD after an abortion for a gestational age between 12 weeks zero days and 23 weeks 6 days. Immediate insertions occur during the visit for the abortion immediately after the abortion is complete, interval insertions will be scheduled for not earlier than two weeks and not later than four weeks after the abortion.
  Arms: 2

SUMMARY:
Hypothesis

Intrauterine contraception placed immediately after a second trimester abortion will result in fewer pregnancies than current standard practice of intended placement at 4 weeks post-abortion.

Study Design

Randomized Controlled Trial after their second trimester abortion comparing immediate with delayed insertion of IUC, and a non intervention control group choosing non-intrauterine contraception. Participants choosing an IUC will be randomly assigned to immediate or delayed insertion. The investigators primary outcome is pregnancy rate within one year.

DETAILED DESCRIPTION:
This Randomized Controlled Trial will be offered to women choosing to have a LNG-IUC or CuT380 after an abortion for gestational ages from 12 to 24 weeks. [delete next insert]"and a non intervention control group offered to all others having abortions at this gestational age". Participants choosing an LNG-IUC or CUT380 will be randomly assigned to immediate or interval insertion. In conjunction with follow up visits and questionnaires, the British Columbia Linked Health Database access will determine pregnancy rate within one year for the two intervention groups [delete next insert] and in relation to the various contraceptive choices made by the women not choosing intrauterine contraception. All women will complete surveys at 3, 6, 12, 24, 36, 48 and 72 months on their satisfaction with the contraceptive method chosen and on their satisfaction with study participation.

ELIGIBILITY:
Inclusion Criteria:

1. Have completed informed consent for an abortion at gestation between 12 weeks zero days and 23 weeks 6 days, and
2. Choosing an IUC (either LNG-IUC or CuT380-IUC) for contraception post abortion, and
3. Residents of British Columbia, registered with the Medical Services Plan health care system.

Exclusion Criteria:

1. Intention to move from BC within the next year
2. Intention to conceive within the next year.
3. Any of the following contraindications to use of a LNG-IUC or a CuT380-IUC
4. Post Randomization Exclusion:

uterine perforation at the time of abortion

bleeding of more than 500 cc during abortion

any of the above exclusions detected at time of abortion

Min Age: 10 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2009-06; Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate at one year | 12 months
  The one year pregnancy rate outcome will be determined using a pragmatic approximation based on the varying exactitude of imputations based on provincial Medical Service Plan billings related to abortions, miscarriages, still births and live births. Subsequent abortions performed within our study clinics for enrolled participants will be noted along with specific clinical information on pregnancy duration. For abortions performed elsewhere such as those for BC university students studying out of province, or those performed by individual physicians at rural or remote hospitals within BC, exact gestation may not be available. In the BC health administrative databases abortions are billed as under 7 weeks for medical abortions, and as under 14 weeks, 14 weeks to under 18 weeks, and 18 weeks and over for surgical abortions. Miscarriages by definition occur anytime under 20 weeks or are classed as still birth when over 20 weeks of gestation.

SECONDARY OUTCOMES:
Rates at one year for Expulsion, Continuation of use, Satisfaction with method, Adverse events. | 60 months
  Secondary outcomes will be assessed initially at one year, then annually through the five year device effectiveness period.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy V. Norman, Ph.D, Principal Investigator — University of British Columbia; Brian Fitzsimmons, MD, Study Director — University of British Columbia; Lyda Dicus, Study Chair — University of British Columbia
Locations (3):
- Canada (3):
  - Kelowna General Hospital Women's Services Clinic, Kelowna, British Columbia
  - BC Women's Hospital, Vancouver, British Columbia
  - Elizabeth Bagshaw Women's Clinic, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No